CLINICAL TRIAL: NCT04722770
Title: Clinical Development and Evaluation of a Deep Learning Approach to Improve Diagnostic Accuracy
Brief Title: Clinical Development of Deep Learning for the OtoSight
Status: Completed | Type: Observational
Sponsor: PhotoniCare, Inc. (Industry)
Collaborators: University of Pittsburgh (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 000002; R44DC017422 (NIH)
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-05

CONDITIONS: Otitis Media Acute
Keywords: Ear Infection; Otitis Media; Otitis Media with Effusion; Machine Learning
MeSH Terms: conditions — Otitis Media; Otitis; Otitis Media with Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Pediatric patients with possible ear infections: Pediatric patients presenting with otitis media (acute otitis media or otitis media with effusion) will be imaged with the PhotoniCare OtoSight.
  Interventions: Device: PhotoniCare OtoSight Middle Ear Scope

INTERVENTIONS:
Device: PhotoniCare OtoSight Middle Ear Scope — PhotoniCare OtoSight imaging using a near-infrared laser

SUMMARY:
The objective of this study is to clinically develop and evaluate a machine learning approach to improve the performance and data interpretation of the PhotoniCare OtoSight Middle Ear Scope in pediatric patients presenting at the primary care office for suspected ear infections. In this observational study, results of OtoSight imaging will not affect patient standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients presenting for an office visit with ear-related complaints

Exclusion Criteria:

* Otoscopy contra-indicated or not possible per attending clinician's decision, Down's syndrome (due to abnormalities in ear canal anatomy)

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children presenting to the pediatric clinic with suspected ear infection
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
PhotoniCare OtoSight imaging exam | 1-5 minutes; at first and only study visit
  Optical coherence tomography imaging to evaluate the middle ear.

SECONDARY OUTCOMES:
Adverse events | 15-30 minutes; at first and only study visit
  Rate of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Shelton, PhD, Principal Investigator — PhotoniCare, Inc.
Locations (1):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No